CLINICAL TRIAL: NCT04665258
Title: Corona Virus Disease 19 (COVID-19) Vaccine and Impact on Fertility Study
Brief Title: Male Reproduction COVID Sequelae Study (MARCOS).
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit participants
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Associate Professor, University of Miami
Other Study IDs: 20201451
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Infertility, Male
Keywords: COVID-19 Vaccine
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 vaccine group: Participants scheduled to receive the COVID-19 vaccine will be evaluated on its effect on semen parameters for up to 6 months post vaccination.

SUMMARY:
The purpose of this study is to investigate the effects of COVID-19 Vaccination on semen parameters and to determine how long these possible changes may last following vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving COVID-19 vaccines
2. Male age 18-50 years old

Exclusion Criteria:

1. Adults unable to consent
2. Women
3. Prisoners
4. Men who have been receiving Testosterone replacement therapy or anabolic steroids within the last year
5. Men with a history of Azoospermia
6. Men with a genetic or other medical condition known to be associated with decreased semen parameters (i.e. Klinefelter's syndrome, Y-Chromosome Microdeletion (YCMD), post-chemotherapy treatment, etc.)
7. Positive COVID-19 test within the last 3 weeks

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young men of reproductive age scheduled for COVID-19 Vaccine
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Sperm concentration | up to 6 months
  As measured from semen samples.
Sperm motility | up to 6 months
  As measured from semen samples.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No